CLINICAL TRIAL: NCT00219895
Title: Assessment of Induced Sputum as a Tool to Evaluate Anti-Inflammatory Agents in Patients With Cystic Fibrosis
Brief Title: Assessment of Inflammatory Mediators (AIM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramsey, Bonnie, MD (Individual)
Collaborators: Cystic Fibrosis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFOM0003
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2007-12-25 (Estimated); Status verified 2006-08

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Anti-inflammatory Agents; Ibuprofen
MeSH Terms: conditions — Cystic Fibrosis | interventions — Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen

SUMMARY:
Specific Aim: To determine whether neutrophils, active elastase, and cytokines measured in sputum induced using hypertonic saline are useful screening tests for determining if a particular agent with known anti-inflammatory properties is a suitable candidate for more extensive clinical trials in patients with CF. This aim will be addressed using an anti-inflammatory agent, ibuprofen, that has been shown to have clinical benefit in CF. A "no treatment" arm will be included as the control group.

DETAILED DESCRIPTION:
Inflammation clearly contributes to the progression of cystic fibrosis (CF) lung disease. Anti-inflammatory therapy with alternate-day corticosteroids and twice-daily high-dose ibuprofen in patients with CF has shown clinical benefit, but adverse effects and other considerations have markedly limited their use. Therefore, alternative anti-inflammatory agents are urgently needed. Results from the clinical trials of alternate-day corticosteroids and high-dose ibuprofen in CF indicate that anti-inflammatory therapy will probably not result in improvement in pulmonary function, but will slow the rate of decline. This expectation imposes constraints on the design of studies to test new anti-inflammatory agents, requiring that they use many patients over a considerable period of time (years, rather than the months that are necessary to evaluate anti-infective or anti-obstructive therapies). Thus, it is highly desirable to design a strategy for evaluation of prospective anti-inflammatory agents that will allow for the selection of only the most promising agents for further study in Phase III type trials. Of additional concern is the fact that some pharmaceutical firms have not pursued development of anti-inflammatory agents for CF because there were no early indicators of efficacy. This presents an insurmountable hurdle for translation of research advances into clinical treatments. Some means of screening candidate drugs is urgently required. This study will assess the measurement of inflammatory mediators in induced sputum as one such strategy. The hypothesis to be tested is that ibuprofen will reduce neutrophils, active elastase, and pro-inflammatory cytokines in induced sputum after 4 weeks of therapy in patients with CF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 10 years of age or older.
* Confirmed diagnosis of CF based on the following criteria:

  * positive sweat chloride >= 60 mEq/liter (by pilocarpine iontophoresis) and/or
  * a genotype with two identifiable mutations consistent with CF, and
  * accompanied by one or more clinical features consistent with the CF phenotype
* FEV1 >= 50% predicted value (subjects >= 10 - <18 years of age) or >= 40% predicted value (subjects >= 18 years of age)
* Clinically stable with no evidence of acute upper or lower respiratory tract infection or current pulmonary exacerbation within the 14 days prior to Visit 1 (Day 0)
* Ability to reproducibly perform spirometry and peak flow measurements
* Ability to understand and sign a written informed consent or assent and comply with the requirements of the study

Exclusion Criteria:

* Use of an investigational agent within the 4-week period prior to Visit 1 (Day 0)
* Chronic daily use of ibuprofen, celecoxib, or other selective COX-2 inhibitors, other NSAIDs, or systemic or inhaled corticosteroids within the 4 weeks prior to Visit 1 (Day 0) or acute usage within 72 hours prior to Visit 1 (Day 0)
* History of hypersensitivity to beta-agonists
* History of hypersensitivity to sulfonamides, aspirin, or other NSAIDs
* Oxygen saturation < 92% on room air at Visit 1 (Day 0)
* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* History of hemoptysis >= 30 cc per episode during the 30 days prior to Visit 1 (Day 0)
* Significant history of hepatic, cardiovascular, renal, neurological, hematologic, or peptic ulcer disease
* SGOT (ALT) or SGPT (AST) > 3 times the upper limit of normal at screening, documented biliary cirrhosis, or portal hypertension
* Creatinine > 1.8 mg/dL at screening
* Inability to swallow pills
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2004-08; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Changes in markers of inflammation in induced sputum samples: total white cell count, total neutrophil count, percent neutrophils, active elastase, and cytokines.

SECONDARY OUTCOMES:
(1) Alterations in laboratory evaluations: CBC, ESR, CRP, serum chemistry profile, urinalysis, and spirometry. (2) Adverse events associated with sputum induction or administration of study medications

CONTACTS AND LOCATIONS:
Overall Officials: James Chmiel, MD, MPH, Principal Investigator — Case Western Reserve University - Rainbow Babies and Children's Hospital
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University - Packard Children's Hospital, Palo Alto, California
  - University of California - San Diego, San Diego, California
  - University of Colorado Health Sciences Center - Children's Hospital, Denver, Colorado
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Harvard University - Children's Hospital of Boston, Pulmonary Division, Boston, Massachusetts
  - University Of Minnesota, Minneapolis, Minnesota
  - Washington University - St. Louis Children's Hospital, St Louis, Missouri
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Baylor College of Medicine - Texas Children's Hospital, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah